CLINICAL TRIAL: NCT05495360
Title: Effect of Omega 3 Enriched Oral Nutritional Supplement on Nutritional Status of CRC and NSCLC Patients
Acronym: OMENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SBB20R&35115
Record Dates: First submitted 2022-08-02; First posted 2022-08-10 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Malnutrition; Oncology
Keywords: Oral nutritional supplement; Oncology; Omega 3
MeSH Terms: conditions — Malnutrition; Neoplasms | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): twice daily serving of the study product
  Interventions: Dietary Supplement: Oral Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: Oral Nutritional Supplement — twice daily serving of the study product

SUMMARY:
A single arm intervention study examining the effect of an omega 3 enriched oral nutritional supplement on nutritional status of CRC and NSCLC patients

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven CRC or histologically or cytologically proven NSCLC
2. Eligible and scheduled for at least 2 cycles of 4-week cycles of systemic treatment, 3 cycles of 3-week cycles of systemic treatment or 4 cycles of 2-week cycles of systemic treatment
3. At risk of malnutrition or malnourished [PG-SGA-SF > 4]
4. Performance status ECOG 0 or 1
5. Weight loss grade 0-3 according to Martin et al1
6. <11% weight loss in the past 6 months
7. Age ≥ 18 years
8. Written informed consent

Exclusion Criteria:

1. Presence of ileostoma or ileal pouch
2. GI-related or major surgery in 30 days prior to baseline
3. Severe hypercalcemia, i.e. total calcium level, corrected for albumin ≥ 14.0 mg/dL (3.5 mmol/L)
4. Use of ONS, enteral nutrition or parenteral nutrition within 14 days prior to entry into the study
5. Use of fish oil containing supplements, within 30 days prior to entry into the study or expected to use this during the study
6. Use of more than 200 iU/day of vitamin D containing supplements within 30 days prior to entry into the study or expected to use this during the study
7. Life expectancy of < 3 months
8. Severe renal dysfunction (<29 ml/min/1.73m2 eGRF or albumin:creatinine (ACR) > 30) or hepatic encephalopathy
9. Allergy to cow's milk protein or fish, known protein sensitivity or suffering galactosemia
10. Known pregnancy or lactation
11. Current alcohol or drug abuse in opinion of the investigator
12. Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements
13. Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Change in EPA concentration in the phospholipid fraction of the erythrocyte membrane [% of total fatty acids] | at end of first in-study treatment cycle compared to baseline

SECONDARY OUTCOMES:
Change in protein intake [g/day] [key secondary outcome) | at end of first in-study treatment cycle compared to baseline
Change in protein intake [g/kg bw/day] [key secondary outcome) | at end of first in-study treatment cycle compared to baseline
Change in energy intake [kcal/day] | at end of first in-study treatment cycle compared to baseline
Change in energy intake [kcal/kg bw/day] | at end of first in-study treatment cycle compared to baseline
Provided vitamin D supplementation [µg/day] by the test product | Throughout total intervention period - about 2 months
Change in fatty acid profile in the phospholipid fraction of the cell membrane of erythrocytes [% of total fatty acids] | at end of first in-study treatment cycle compared to baseline

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Brussels
  - AZ Delta, Roeselare
- Czechia (2):
  - Faculty Hospital Brno, Brno
  - Fakultní nemocnice Bulovka, Prague
- Cork University Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No